CLINICAL TRIAL: NCT00211718
Title: Intra-Articular Injection of Botulinum Toxin Type A for the Treatment of Shoulder Pain: A Randomized, Double Blinded, Placebo Controlled Trial
Brief Title: Intra-Articular Injection of Botulinum Toxin Type A for Shoulder Pain
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Minneapolis Veterans Affairs Medical Center (U.S. Federal Agency)
Collaborators: Allergan (Industry); Center for Veterans Research and Education (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB Protocol Number 03404B
Record Dates: First submitted 2005-09-14; First posted 2005-09-21 (Estimated); Last update posted 2005-11-03 (Estimated); Status verified 2005-08

CONDITIONS: Arthritis; Shoulder Pain
Keywords: shoulder pain; arthritis; intra-articular botulinum toxin a; joint pain
MeSH Terms: conditions — Arthritis; Shoulder Pain; Arthralgia | interventions — Botulinum Toxins, Type A

INTERVENTIONS:
Drug: intra-articular botulinum toxin type a

SUMMARY:
The purpose of this study is to determine whether intra-articular botulinum toxin type A is effective in the treatment of chronic joint pain.

DETAILED DESCRIPTION:
Chronic shoulder pain unresponsive to oral medications and intra-articular corticosteroids is an important treatment problem, especially for the young, very old and those with complex medical problems that preclude joint reconstructive surgery. We hypothesized that intra-articular botulinum toxin could provide important joint pain relief in these patients. This is a prospective, double blined, placebo controlled 6month trial with an open label extension phase when pain returns to baseline levels (re-injection with 100units of botulinum toxin and 6 months followup thereafter).

Comparisons: Intra-articular injection of botulinum toxin type a will be compared to intra-articular injection of placebo ( lidocaine then saline).

ELIGIBILITY:
Inclusion Criteria:

* • Male or female subjects, 18 years of age or older.

  * Written informed consent and written authorization for use or release of health and research study information have been obtained.
  * Subject has chronic Shoulder joint pain for more than 1 year.
  * Subject has pain >4.5 on numerical rating scale of 0 to 10.
  * Ability to follow study instructions and likely to complete all required visits.
  * Negative urine pregnancy test on the day of treatment prior to the administration of study medication (for females of childbearing potential if applicable)
  * Patients previously treated with intra-articular corticosteroid or viscosupplementation injections.
  * Patients with rheumatoid arthritis must have failed therapy with standard DMARDs (disease modifying anti-rheumatic drugs) and anti-TNF agents unless they have a contraindication to TNF blockers.
  * Patients who were considered not to be candidates for Shoulder joint replacement because of young age, abnormalities in periarticular tissues or because of co-morbid conditions.
  * Must be ambulatory and able to perform sit to stand.

Exclusion Criteria:

* Use of aminoglycoside antibiotics, curare-like agents, or other agents that might interfere with neuromuscular function.
* Any medical condition that may put the subject at increased risk with exposure to botulinum neurotoxin including diagnosed myasthenia gravis, Eaton-Lambert syndrome, amytrophic lateral sclerosis, any other disorder that might interfere with neuromuscular function or the presence of severe peripheral neuropathy.
* Females who are pregnant, breast-feeding, or planning a pregnancy during the study or who think that they may be pregnant at the start of the study, or females of childbearing potential who are unable or unwilling to use a reliable form of contraception during the study.
* Known allergy or sensitivity to any of the components in the study medication.
* Evidence of recent alcohol or drug abuse.
* Infection at injection site or systemic infection (postpone study entry until one week following recovery.
* Known, uncontrolled serious systemic disease and/or life expectancy less than 12 months.
* Concurrent participation in another investigational drug or device study or participation in the 30 days immediately prior to study enrollment.
* Any condition or situation that, in the investigator's opinion, may put the subject at significant risk, confound the study results, or interfere significantly with the subject's participation in the study.
* Patients whose pain is rated as less than 4.5 on a 10 point Numerical Pain Rating scale at the screening visit
* Patients on coumadin or heparin because of increased risk of bleeding in the joint
* Serious or unstable psychiatric disease or cognitive impairment that would limit evaluation of response to treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2004-07; Study Completion 2007-06

PRIMARY OUTCOMES:
: Primary Outcomes:
Change in Pain Score
Change in Joint Function
Patient Global Assessment

SECONDARY OUTCOMES:
Secondary Outcomes:
Pain Relief
Change in Health Status Quality of Life-SF36
Change in Disease specific Health Related QOL-WOOS
Function improvement - Range of Motion, SPADI, Simple Shoulder tes
Physican Assessment of Pain and Global Assessment of Improvement
Safety Measure,

CONTACTS AND LOCATIONS:
Overall Officials: Maren L Mahowald, MD, Principal Investigator — Minneapolis VAMC
Locations (1):
- Minneapolis VAMC, Minneapolis, Minnesota, United States